CLINICAL TRIAL: NCT03587402
Title: Effects of Transcutaneous Perineal Stimulation Versus Anal Stimulation on Urinary Incontinence After Radical Prostatectomy
Brief Title: Effects of Transcutaneous Perineal Stimulation Versus Anal Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAPbarcelona (Other)
Responsible Party: Principal Investigator, Regina Pané Alemany, Principal investigator, RAPbarcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAP47747176G
Record Dates: First submitted 2018-06-27; First posted 2018-07-16 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Urinary Incontinence; Radical Prostatectomy; Pelvic Floor
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous perineal stimulation (Experimental): Patient is asked to lie down with legs slightly bend and two adhesive electrodes are attached transcutaneous on base of penis and on perineum. Stimulation current is administrated half time with a fixed frequency of 30 Hz and half time with 50 Hz. Pulse increased until the patient perceives the current. Sessions lasted for 30 minutes weekly for 10 weeks.
  Interventions: Other: Transcutaneous perineal stimulation
- Anal stimulation (Active Comparator): Patient is asked to lie down with legs slightly bend and an electrical probe is inserted into the anus. Stimulation current is administrated half time with a fixed frequency of 30 Hz and half time with 50 Hz. Pulse increased until the patient perceives the current. Sessions lasted for 30 minutes weekly for 10 weeks.
  Interventions: Other: Anal stimulation

INTERVENTIONS:
Other: Transcutaneous perineal stimulation — Surface stimulation
  Arms: Transcutaneous perineal stimulation
Other: Anal stimulation — Intra-cavitary stimulation
  Arms: Anal stimulation

SUMMARY:
This study evaluates whether surface perineal stimulation is as effective as anal stimulation in reducing urinary incontinence secondary to radical prostatectomy.

Half of participants will receive a treatment with surface perineal stimulation, while the other half will receive a treatment with anal stimulation.

DETAILED DESCRIPTION:
Pelvic floor muscle training is the most common non-invasive intervention for urinary incontinence secondary to radical prostatectomy. Perineal stimulation has a significant positive impact on the early recovery of urinary continence after this intervention.

The perineal stimulation can be applied with surface electrodes or with an intra-cavitary probe placed in the anus. The two techniques are commonly used. Each techniques stimulates different anatomical points of perineum, and it is a question if both have the same effectiveness or, one of the two techniques has greater effect than the other.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone a radical prostatectomy surgical procedure.
* Presenting involuntary urine losses after radical prostatectomy intervention. (IU grade I, II or III)
* Do not exceed the year since the surgical intervention.
* Accept to participate in the study and grant signed informed consent.

Exclusion Criteria:

* Follow a pharmacological treatment for the UI.
* Presenting anatomical malformations of the pelvic floor musculature.
* Carry pacemaker.
* Present anal fistulas.
* suffer from serious psychic disorders.
* Presenting lower urinary tract infections.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As it is a prostatic pathology, only men participate in the study
Enrollment: 70 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Effects of transcutaneous perineal stimulation compared to anal stimulation | Baseline, 6 and 10 weeks
  A change of the urine grams last in 24 hours

SECONDARY OUTCOMES:
Asses quality of life | Baseline and 10 weeks
  Asses the perceived quality of life of patients in the study. It will be evaluated with the questionnaire I-QOL. It measures the effect of urinary incontinence on quality of life.
  The I-QOL have 22 items and is divided into 3 subscales: avoidance and limiting behavior, psychosocial impact, social embarrassment. More puntuation means more quality of life.
Assess adverse effects | 10 weeks
  Identify adverse effects for each of the treatments

CONTACTS AND LOCATIONS:
Overall Officials: Regina Pané, Principal Investigator — RAPbarcelona; Inés Ramírez, Study Director — RAPbarcelona
Locations (1):
- Regina Pané Alemany, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pane-Alemany R, Ramirez-Garcia I, Carralero-Martinez A, Blanco-Ratto L, Kauffmann S, Sanchez E. Efficacy of transcutaneous perineal electrostimulation versus intracavitary anal electrostimulation in the treatment of urinary incontinence after a radical prostatectomy: randomized controlled trial study protocol. BMC Urol. 2021 Jan 28;21(1):12. doi: 10.1186/s12894-020-00718-y. PMID 33509164